CLINICAL TRIAL: NCT03922295
Title: Endoscopic Tympanoplasty: Single Versus Double Flap Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha A.Elkholy, ORL-HNS Resident, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1ORL
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic double flap group (Active Comparator)
  Interventions: Procedure: Endoscopic tympanoplasty
- endoscopic single flap group (Active Comparator)
  Interventions: Procedure: Endoscopic tympanoplasty

INTERVENTIONS:
Procedure: Endoscopic tympanoplasty — In the double flap group, graft is placed via elevation of both posterior and anterior flaps.
  In the single flap group, graft is placed via elevation of posterior flap only

SUMMARY:
Aim of this study is to compare results of double and single flap techniques for tympanoplasty in chronic suppurative otitis media patients. Inclusion criteria include total or subtotal tympanic membrane perforations with limited anterior remnant and should be dry for at least 3 months. Patients with persistent discharge, cholesteatoma, ossicular affection or those with recurrent perforations after previous myringoplasty were excluded. Also, patients with uncontrolled diabetes, chronic liver and kidney diseases and immuno-compromised patients are not included in this study. Patients are divided into two groups, endoscopic double flap group and endoscopic single flap group. Healing and hearing outcomes were evaluated 3 months postoperative. Also, post-operative pain scores and complications were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic suppurative otitis media with total or subtotal tympanic membrane perforation with limited anterior remnant.
* dry perforation for at least 3 months.

Exclusion Criteria:

* Recurrent perforation after previous myringoplasty.
* Ossicular disruption or fixation.
* immune-compromised patients including uncontrolled diabetics, chronic liver and kidney diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Healing or graft take rate | 3 months after surgery
  closure of tympanic membrane perforation

CONTACTS AND LOCATIONS:
Overall Officials: Noha A Elkholy, Principal Investigator — ORL-HNS department, Faculty of Medicine, Mansoura University; Mohammed A Salem, Study Director — ORL-HNS department, Faculty of Medicine, Mansoura University; Abdelwahab M Rakha, Study Chair — ORL-HNS department, Faculty of Medicine, Mansoura University
Locations (1):
- ORL-HNS department,Mansoura University Hospital, Faculty of Medicine, Mansoura University, Al Mansurah, ElDakahlia, Egypt

REFERENCES:
- [Derived] El-Kholy NA, Salem MA, Rakha AM. Endoscopic single versus double flap tympanoplasty: a randomized clinical trial. Eur Arch Otorhinolaryngol. 2021 May;278(5):1395-1401. doi: 10.1007/s00405-020-06212-3. Epub 2020 Jul 20. PMID 32691232

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03922295/Prot_SAP_000.pdf